CLINICAL TRIAL: NCT01448655
Title: Prospective Epidemiological Study to Expand Knowledge on Efficacy and Safety of a Routine Post-operative Supportive Therapy With the Mistletoe Extract Iscador® Qu Within Oncological Treatment of Colorectal Cancer Stages UICC II-IV
Brief Title: Iscador Qu as Supportive Treatment in Colorectal Cancer (Union International Cancer Control, UICC Stages II-IV)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IFAG AG (Industry)
Collaborators: Hiscia Society for Cancer Research (Unknown); IFAG Basel AG (CRO), both Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: ISC-4.1.5; 2010-018682-31 (EudraCT Number)
Record Dates: First submitted 2011-03-29; First posted 2011-10-07 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; mistletoe; supportive treatment; long-term study; non-interventional cohort study; controlled study with parallel groups
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test group with Iscador® Qu: The test group will receive the mistletoe extract Iscador® Qu as supportive treatment in addition to post-operative conventional oncological therapy (radio-, chemo-, targeted therapy).
- Control group: The parallel control group will receive no mistletoe but only post-operative conventional oncological therapy (radio-, chemo-, targeted therapy).

SUMMARY:
Efficacy and safety of a supportive treatment with European mistletoe extract Iscador® Qu ("quercus", i.e. from oak tree) in patients with colorectal cancer (Union for International Cancer Control, UICC stages II-IV), in addition to post-operative conventional oncological therapy (radio-, chemo-, targeted therapy) as compared to a parallel group with conventional therapy only.

Primary Endpoints: Reduction of adverse effects of conventional therapy; reduction of therapy or disease induced symptoms (both are quality of life parameters and evaluated after 1 year); prolongation of disease free and/or overall survival (DFS, OS) after 5 years.

Prospective observational confirmation study of previous retrospective cohort study.

As this is a non-interventional cohort study, all therapies and measurements are performed on directive by the treating physician and/or request by the patient only.

DETAILED DESCRIPTION:
see summary

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of colorectal cancer, UICC stage II-IV
* Age between 18 (Austria: 19) and 85 years
* No previous malign tumor
* Surgical resection of the tumor if indicated
* (Post-operative) conventional oncological therapy and measurements, or passive after-care ("best care")
* Follow-up for several years feasible
* Patient gives written consent to use the anonymized date for evaluation

Exclusion Criteria:

* Anal cancer
* Other Iscador® sorts than Qu in the test group
* Other mistletoe preparations in the test group
* Any mistletoe preparation in the control group
* Non-oncological immunomodulating, -stimulating or -suppressive drugs (e.g. Echinacea, interferons, Polyerga®, BCG, azathioprine). Allowed are approved tumor inhibiting immuno- or targeted therapies (e.g. bevacizumab, cetuximab) and tumor specific vaccines
* HIV infection, Aids, organ transplantation
* High-dose systemic glucocorticoids
* Contraindications for Iscador® Qu (allergy against mistletoe, acute inflammatory disease or fever > 38.5°C, active tuberculosis, hyperthyreosis with not-adjusted metabolism, primary brain or spinal tumor, brain metastases)
* Known mistletoe intolerance
* Patients participating in another clinical study with non-approved substances

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients visiting the center with colorectal cancer stage UICC II-IV and meeting the eligibility criteria will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time (DFS). | 5 years

SECONDARY OUTCOMES:
Number of patients with at least one therapy or disease induced symptom (surrogate parameter for quality of life) | 1 year
  As key symptom, the fatigue syndrome will be evaluated separately.
Mean values of Karnofsky performance status, Eastern Cooperative Oncology Group (ECOG) score | 1 year
Interim analysis on overall survival time (OS) in UICC stage IV patients | 2 years
Safety of Iscador® Qu (number of patients with systemic or local adverse events (AE) to Iscador® Qu) | 5 years
  Adverse events (local and/or systemic) contributable to Iscador® Qu
Number of patients with unexpected adverse events (UAE) contributed to conventional oncological therapy (radio-, chemo-, targeted therapy). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof. M.D., Principal Investigator — University Clinic Halle (Saale)
Locations (9):
- Austria (2):
  - 5th Med., Clinic Hietzing, Vienna
  - University Vienna, Vienna
- Germany (7):
  - Augusta Clinic, Bochum
  - MVZ Fulda, Fulda
  - University Clinic - Internal Medicine I, Halle
  - Hospital Herdecke, private University, Herdecke
  - Med. Clinic III, University Munich, Grosshadern, Munich
  - Clinic Kloster Paradiese, Soest
  - Med 1, University Clinic Ulm, Ulm

REFERENCES:
- [Background] Ostermann T, Raak C, Bussing A. Survival of cancer patients treated with mistletoe extract (Iscador): a systematic literature review. BMC Cancer. 2009 Dec 18;9:451. doi: 10.1186/1471-2407-9-451. PMID 20021637
- [Background] Friedel WE, Matthes H, Bock PR, Zanker KS. Systematic evaluation of the clinical effects of supportive mistletoe treatment within chemo- and/or radiotherapy protocols and long-term mistletoe application in nonmetastatic colorectal carcinoma: multicenter, controlled, observational cohort study. J Soc Integr Oncol. 2009 Fall;7(4):137-45. PMID 19883529
- [Background] Ziegler R. Mistletoe Preparation Iscador: Are there Methodological Concerns with Respect to Controlled Clinical Trials? Evid Based Complement Alternat Med. 2009 Mar;6(1):19-30. doi: 10.1093/ecam/nem121. Epub 2007 Oct 4. PMID 18955241